CLINICAL TRIAL: NCT06594471
Title: Comprehensive Assessment of Characteristics and Outcomes of Gemelli Adolescents and Young Adults Diagnosed With Gynecological Cancer
Brief Title: Comprehensive Assessment of Clinical Characteristics and Outcomes of Gemelli Adolescents and Young Adults
Acronym: G-AYA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 6432
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire on late-term physical effects — Patients will be asked to indicate any potential late-term physical effects following cancer treatment: neurocognitive, auditory, ocular, oral/dental, dermatologic, cardiovascular, pulmonary, gastro-intestinal, urinary tract, genital, endocrine/metabolic, musculoskeletal, neurological, immune disorders and occurrence of any subsequent malignant neoplasms.
Other: Questionnaire on sexual and reproductive health outcomes — Patients will be asked to complete the following questionnaires: Body Appreciation Scale-2 (BAS-2), Body Image Scale (BIS), EORTC QLQ-SH22, Body Image Scale in Gynecological Cancer (SABIS-G). Patients who underwent a fertility-sparing procedure will be asked to fill out the Reproductive Concerns after Cancer (RCAC) and Decision Regret Scale (DRS), whereas those who experienced iatrogenic menopause will complete the MENQOL questionnaire to assess menopause-related quality of life.
Other: Questionnaire on psychological outcomes — Patients will be asked to complete the following questionaires: EORTC QLQ-C30, Clinical outcomes in Routine Evaluation (CORE-OM), Ten Item Personality Inventory (TIPI), Hospital Anxiety and Depression Scale (HADS), General Self-Efficacy (GSE) Scale, Mini-Mental Adjustment to Cancer (Mini-MAC), Cancer Worry Scale (CWS), Multidimensional Scale of Perceived Social Support (MSPSS), the Patient Health Engagement scale and the Supportive Care Needs Survey-Short Form (SCNS-SF34).
Other: Questionnaire on social outcomes — Patients will be asked to complete the following questionaires: Medical Consumption Questionnaire (iMCQ), Productivity Cost Questionnaire (iPCQ) and the Comprehensive Score for Financial Toxicity - Functional Assessment of Chronic Illness Therapy (COST-FACIT) questionnaire.

SUMMARY:
The Adolescent and Young Adults cancer population encompass patients diagnosed with oncological disease at the age of 15-39 years. Although 86% of these patients become long-term cancer survivors, studies have shown that these survival rates lag behind to those of younger and older patients. The underlying reason for this discrepancy is, however, yet poorly understood. Furthermore, these patients may be more often confronted with late effects due to their disease and/or anticancer treatment. Knowledge on Adolescent and Young Adults diagnosed with gynecological cancer at the Fondazione Policlinico Universitario Agostino Gemelli IRCCS hospital in Rome, Italy, is currently lacking and is needed to deliver these patients the best possible care, tailored to their disease characteristics and specific needs.

The primary objective of this monocenter observational study is to determine the number of Gemelli Adolescent and Young Adults diagnosed with gynecological cancer and their clinical characteristics. Secondary objectives will be to determine their oncological, late-term physical effects, sexual and reproductive health, psychological and social outcomes. Tertiary outcomes will be to compare the clinical characteristics and oncological outcomes of Gemelli Adolescents and Young Adults to patients beyond this age-specific cohort who have been treated during the same study period.

DETAILED DESCRIPTION:
Clinical, diagnosis and treatment characteristics will be determined. In addition, oncological (e.g., disease-free and overall survival), late-term physical (e.g., cardiovascular, second primary tumor), sexual and reproductive health (e.g., body image, sexual functioning, fertility preservation, pregnancy rate, premature ovarian insufficiency), psychological (e.g., anxiety and depression) and social (e.g. (un)employment, financial toxicity) outcomes will be determined.

ELIGIBILITY:
Inclusion Criteria:

Gynecological cancer types include but are not limited to the following:

* Ovarian cancer - borderline tumors with invasive peritoneal implants, epithelial carcinoma (endometrioid, clear cell, high-grade serous, low-grade serous, mucinous, undifferentiated), germ cell tumor (dysgerminoma, immature teratomas, yolk sac tumors, embryonal carcinomas, carcinoid tumors), sex cord stromal tumor (gynandroblastoma, granulosa cell tumor, Sertoli-Leydig cell tumor, steroid cell tumor)
* Cervical cancer - squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma, carcinoma in situ with stromal microinvasion (to be considered as microinvasive carcinoma), other
* Endometrial cancer - endometrioid, papillary serous, clear cell, carcinosarcoma
* Sarcoma - uterine sarcoma (incl. leiomyosarcoma, endometrial stromal sarcoma, adenosarcoma)
* Gestational trophoblastic neoplasms - invasive mole, choriosarcoma, placental site trophoblastic tumor, epithelioid trophoblastic tumor, other
* Vulvar-vaginal cancer - squamous cell carcinoma, M. Paget, other

Exclusion Criteria:

1. Mentally disabled or patients with significantly altered mental status that would prohibit understanding and giving informed consent
2. Patients who do not provide informed consent on data collection and storage for scientific purposes

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be included who are diagnosed with gynecological cancer of any tumor type at the age of 15-39 years and have been treated at the Fondazione Policlinico Universitario Agostino Gemelli IRCCS hospital in Rome, Italy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2039-09-30 (Estimated); Study Completion 2040-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes | 10 years
  The number of Adolescents and Young Adults diagnosed with gynecological cancer who receive treatment at the Fondazione Policlinico Universitario Agostino Gemelli IRCCS hospital during a five-year period and their clinical characteristics, i.e., demographics, diagnosis, imaging, treatment and clinical trial participation.

SECONDARY OUTCOMES:
Survival outcomes | 10 years
  Oncological outcomes, i.e., progression-free survival, disease-specific and overall survival
Late-term physical effects - neurocognitive disorders | 10 years
  Number of patients who developed neurocognitive disorders
Late-term physical effects - auditory disorders | 10 years
  Number of patients who developed auditory disorders
Late-term physical effects - ocular disorders | 10 years
  Number of patients who developed ocular disorders
Late-term physical effects - oral/dental disorders | 10 years
  Number of patients who developed oral/dental disorders
Late-term physical effects - dermatological disorders | 10 years
  Number of patients who developed dermatological disorders
Late-term physical effects - cardiovascular disorders | 10 years
  Number of patients who developed cardiovascular disorders
Late-term physical effects - pulmonary disorders | 10 years
  Number of patients who developed pulmonary disorders
Late-term physical effects - gastro-intestinal disorders | 10 years
  Number of patients who developed gastro-intestinal disorders
Late-term physical effects - urinary tract disorders | 10 years
  Number of patients who developed urinary tract disorders
Late-term physical effects - genital disorders | 10 years
  Number of patients who developed genital disorders
Late-term physical effects - endocrine/metabolic disorders | 10 years
  Number of patients who developed endocrine/metabolic disorders
Late-term physical effects - musculoskeletal disorders | 10 years
  Number of patients who developed musculoskeletal disorders
Late-term physical effects - neurological disorders | 10 years
  Number of patients who developed neurological disorders
Late-term physical effects - immune disorders | 10 years
  Number of patients who developed immune disorders
Late-term physical effects - subsequent malignant neoplasms | 10 years
  Number of patients who developed subsequent malignant neoplasms
Sexual outcomes - Body Appreciation Scale-2 | 10 years
  The 10-item BAS-2 uses a 5-point Likert scale with responses ranging from 1 (never) to 5 (always) and has demonstrated positive ties between body appreciation and one's psychological well-being (e.g., self-esteem, optimism, positive affect, and negative links with body surveillance, body shame, and body dissatisfaction)
Sexual outcomes - Sexual Adjustment and Body Image Scale in Gynecological cancer (SABIS-G) | 10 years
  The Sexuality and Body Image Scale for women with Gynecological cancer (SABIS-G) consists of a 7-item measure with 3 items related to body image and 4 related to sexual adjustment. To score the SABIS-G each variable is scored from 1 to 5, with 5 as the best outcome. The body image subscale sum ranges from 3 to 15 and the sexual adjustment subscale sum ranges from 4 to 20.
Sexual outcomes - Female Sexual Function Index (FSFI) | 10 years
  The Female Sexual Function Index (FSFI) is a survey measuring the sexual functioning of women in six different domains: desire, arousal, lubrication, orgasm, satisfaction and pain over the past 30 days. Each domain is scored from 0 to 5 with 5 as the best outcome.
Sexual outcomes - EORTC Sexual Health (SH-22) questionnaire | 10 years
  The 22-item EORTC sexual health questionnaire developed to assess sexual health in male and female cancer patients and cancer survivors and ranges from 1 to 4 with 4 as the best outcome.
Reproductive outcomes - fertility preservation | 10 years
  Number of patients who underwent fertility preservation, number of pregnancies achieved, number of live births achieved
Reproductive outcomes - Decision Regret Scale (DRS) | 10 years
  The Decision Regret Scale (DRS) measures distress or 'remorse' after a health care decision and ranges from 1 to 5 with 5 as the worst outcome
Reproductive outcomes - Reproductive Concerns After Cancer (RCAC) scale | 10 years
  The Reproductive Concerns After Cancer (RCAC) scale is a multidimensional measure of possible reproductive concerns of women following cancer diagnosis and treatment, yielding six subscale scores: fertility potential, partner disclosure of fertility status, child's health, personal health, acceptance of possible infertility, and becoming pregnant. The scale ranges from 1 to 5 with 5 as the worst outcome.
Reproductive outcomes - Iatrogenic menopause | 10 years
  Type of treatments received related to iatrogenic menopause
Reproductive outcomes - Menopause Quality of Life (MenQoL) questionnaire | 10 years
  The extent of menopause-related disturbances patients experienced, ranging from 0 to 6 with 6 as the worst outcome.
Psychological outcomes - EORTC-C30 general quality of life questionnaire | 10 years
  This is a 30-item HRQoL questionnaire consisting of five functional scales (physical, role, cognitive, emotional, and social), a global quality-of-life scale, three symptom scales (fatigue, pain, nausea and vomiting) and a number of single items assessing common symptoms (dyspnea, loss of appetite, sleep disturbance, constipation, and diarrhea) and the perceived financial impact of the disease. It has 28 items ranging from 1 to 4 with 4 as the worst outcome and two items ranging from 0 to 7 with 7 as the best outcome.
Psychological outcomes - Clinical outcomes in Routine Evaluation (CORE-OM) | 10 years
  Clinical outcomes in Routine Evaluation (CORE-OM) is a 34-item evaluation covering four domains: wellbeing, problems, functioning and risk. The score ranges from 0 to 4 with 4 as the worst outcome.
Psychological outcomes - Ten Item Personality Inventory (TIPI) | 10 years
  Ten Item Personality Inventory (TIPI) is a 10-item measure of the Big-Five dimensions (extraversion, agreeableness, conscientiousness, emotional stability, openness).
Psychological outcomes - Hospital Anxiety and Depression Scale (HADS) | 10 years
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item scale with 7 items each for assessing symptoms of anxiety and depression, each item ranging from 0 to 3. Summing up this items a final assesment is obtained: 0-7 = Normal, 8-10 = Borderline abnormal (borderline case),11-21 = Abnormal (case).
Psychological outcomes - Distress thermometer | 10 years
  The distress thermometer is one-item measure that assesses the level of distress patients have experienced in the preceding week and uses a 0-10 rating scale.
Psychological outcomes - General Self-Efficacy (GSE) Scale | 10 years
  The General Self-Efficacy (GSE) Scale consists of ten items to examine the patient's problem-solving abilities. The scale ranges from 1 to 4 with 4 as the best outcome.
Psychological outcomes - Mini-Mental Adjustment to Cancer (Mini-MAC) | 10 years
  The Mini-Mental Adjustment to Cancer (Mini-MAC) scale examines the patients' attitudes towards cancer using a 4-point Likert scale.
Psychological outcomes - Cancer Worry Scale (CWS) | 10 years
  The 8-item Cancer Worry Scale (CWS) assesses concerns regarding cancer diagnosis using a 4-point Likert scale with 4 as the worst outcome.
Psychological outcomes - Multidimensional Scale of Perceived Social Support (MSPSS) | 10 years
  The 12-item Multidimensional Scale of Perceived Social Support (MSPSS) examines to what extent the patient has received support from family members, relatives and friends, ranging from 1 to 7 with 7 as the best outcome.
Psychological outcomes - Patient Health Engagement scale | 10 years
  The 5-item Patient Health Engagement scale examines to what extent the patient is able to manage her disease ranging from 0-7 with 7 as the best outcome.
Psychological outcomes - Supportive Care Needs Survey-Short Form (SCNS-SF34) | 10 years
  The Supportive Care Needs Survey-Short Form (SCNS-SF34) is a 34-item, validated measure of cancer-specific perceived needs across five domains: psychological, health systems and information, physical and daily living, patient care and support, and sexuality. Patients rate their level of need for help in the past month, scale ranges from 1 (no need/not applicable) to 5 (high need).
Social outcomes - Medical Consumption Questionnaire (iMCQ) | 10 years
  Number of occurring contacts with health care providers and time off from work for doctors' visits.
Social outcomes - Productivity Cost Questionnaire (iPCQ) | 10 years
  Productivity Cost Questionnaire (iPCQ) will be used to evaluate the impact of disease on the productivity of a person
Social outcomes - Comprehensive Score for Financial Toxicity - Functional Assessment of Chronic Illness Therapy (COST-FACIT) tool | 10 years
  The Comprehensive Score for Financial Toxicity - Functional Assessment of Chronic Illness Therapy (COST-FACIT) tool represents a patient-reported outcome measure that describes the financial distress experienced by cancer patients using a 5-point Likert scale ranging from 0 to 4 with 4 as the worst outcome.

OTHER OUTCOMES:
Comparison of clinical characteristics with patients beyond this age-specific cohort | 10 years
  Comparison of the clinical characteristics (demographics, diagnosis, imaging, treatment and clinical trial participation) of Gemelli Adolescents and Young Adults diagnosed with gynecological cancer to patients beyond this age-specific cohort who have been treated during the same study period
Comparison of oncological outcomes with patients beyond this age-specific cohort | 10 years
  Comparison of progression-free survival, disease-specific and overall survival between Adolescents and Young Adults (15-39 years old at time of diagnosis) versus patients either younger than 15 and/or older than 39 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC GINECOLOGIA ONCOLOGICA, Roma, Italy